CLINICAL TRIAL: NCT00124709
Title: An Investigation of the Safety and Efficacy of Elidel® 1% Cream in Atopic Disease Modification, Assessed in a 3-year Randomized Double-blind Vehicle Controlled Phase to Evaluate Effects on Atopic Dermatitis in Infants, and a 2-3 Year Open-label Phase to Evaluate the Effect of Early Intervention Versus Delayed Intervention With Elidel® on the Incidence of Asthma in Children
Brief Title: Safety and Efficacy of Pimecrolimus Cream 1% in Atopic Disease Modification
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981CUS09
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Results first posted 2011-03-23 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic, dermatitis, asthma, children, modification; Atopic dermatitis/atopy
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Asthma | interventions — pimecrolimus; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Pimecrolimus
  Interventions: Drug: Pimecrolimus
- 2 (Active Comparator): Corticosteroid
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus cream 1 %
  Other Names: Elidel
  Arms: 1
Drug: Corticosteroid — conventional corticosteroid-based treatment
  Arms: 2

SUMMARY:
This study consists of a 3-year double-blind phase during which patients will receive atopic dermatitis (AD) treatment either with pimecrolimus cream 1% long-term management (LTM) or with a conventional corticosteroid-based treatment (1:1 ratio), followed by a 2 to 3-year open-label (OL) phase (all patients receiving pimecrolimus cream 1% LTM). At the end of the double-blind phase, the two treatment groups will be compared with respect to their efficacy in controlling AD; at the end of the OL phase, the incidence of asthma at the age of 6 years will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of atopic dermatitis
* Family history of atopy
* 3 to 18 months of age at baseline
* At least mild atopic dermatitis at baseline (investigator global assessment [IGA] greater or equal to 2)
* Clinical evidence of atopic dermatitis for no longer than 3 months

Exclusion Criteria:

* Diagnosis of or substantial clinical evidence for food or other allergies at baseline

Other protocol related criteria may apply

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1091 (Actual)
Dates: Start 2003-10; Primary Completion 2008-01 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (36):
- United States (36):
  - Alabama Allergy and Asthma Center, Birmingham, Alabama
  - Northwest Arkansas Pediatric Clinic, P.A., Fayetteville, Arkansas
  - The Children's Clinic of Jonesboro, Jonesboro, Arkansas
  - Southern California Research, Mission Viejo, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford Dermatology Clinic and Clinical Trials Dept, Redwood City, California
  - Capital Allergy Respiratory Disease Center, Sacramento, California
  - Children's Hospital San Diego, San Diego, California
  - Allergy and Asthma Medical Group of Diablo Valley, Inc./ Clinical Research Division, Walnut Creek, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Dermatology Associates and Research, Coral Gables, Florida
  - Emerald Coast Clinical Research, Pensacola, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Indiana University Outpatient Clinical Research, Indianapolis, Indiana
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Dermatology Specialists, Louisville, Kentucky
  - Rx R & D, Metarie, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital - Boston, Boston, Massachusetts
  - Dermatology, PLLC, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Central Dermatology, St Louis, Missouri
  - Skin Specialists, P.C., Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center/Dermatology Section, Lebanon, New Hampshire
  - Children's Medical Group, Hopewell Junction, New York
  - Dermatology Associates of St. Luke's - Roosevelt, New York, New York
  - Calcagno Research and Development, Gresham, Oregon
  - Oregon Health Science University - Dermatology Dept., Portland, Oregon
  - The Childrens' Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Texas Children's Hospital, BCM, Houston, Texas
  - Alpine Medical Group, LLC, Salt Lake City, Utah
  - Granger Medical Clinic, West Valley City, Utah
  - Virginia Clinical Research, Norfolk, Virginia
  - Asthma Inc, Seattle, Washington

REFERENCES:
- [Derived] Spergel JM, Boguniewicz M, Schneider L, Hanifin JM, Paller AS, Eichenfield LF. Food Allergy in Infants With Atopic Dermatitis: Limitations of Food-Specific IgE Measurements. Pediatrics. 2015 Dec;136(6):e1530-8. doi: 10.1542/peds.2015-1444. PMID 26598458

RESULTS

PARTICIPANT FLOW:
Groups:
- Pimecrolimus (Elidel) Treatment Group: Pimecrolimus (Elidel) 1% Cream twice a day/topical corticosteroid rescue
- Control Treatment Group: Management with vehicle/topical corticosteroid rescue.
Period: Overall Study
Arm/Group | Pimecrolimus (Elidel) Treatment Group | Control Treatment Group
Started | 546 | 545
Patients Who Received Study Medication | 543 | 544
Completed | 291 (232 Participants entered the OL phase of the study.) | 273 (232 Participants entered the OL phase of the study.)
Not Completed | 255 | 272
Not completed — Randomized but did not take medication | 3 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 5 | 10
Not completed — Protocol Violation | 3 | 5
Not completed — Withdrawal by Subject | 127 | 136
Not completed — Lost to Follow-up | 114 | 120

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimecrolimus (Elidel) Treatment Group | Control Treatment Group | Total
Number analyzed (Participants) | 543 | 544 | 1087
Age Continuous [Mean (Standard Deviation); unit: months] | 7.1 (3.76) | 7.4 (4.06) | 7.3 (3.91)
Age, Customized [Number; unit: Participants]
  Less than 3 months | 1 | 2 | 3
  3 months to Less than 6 months | 230 | 223 | 453
  6 months to Less than 12 months | 231 | 220 | 451
  12 months to Less than or equal to 18 months | 81 | 99 | 180
  Greater than 18 months | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 218 | 412
  Male | 349 | 326 | 675
Parents' Index of Quality of Life - Atopic Dermatitis Score [Mean (Standard Deviation); unit: Scores on PIQoL-AD Scale] — Parents' Index Quality of Life - Atopic Dermatitis (PIQoL-AD) score = (sum of valid items/number of valid items)*28. Scores range from a total possible minimum value of 0 to a maximum value of 28, with a high total overall score indicating poor quality of life.
  Scores on PIQoL-AD Scale | 6.5 (4.73) | 6.9 (4.92) | 6.7 (4.83)

OUTCOME MEASURES:

1. Primary Outcome: Atopic Dermatitis (AD) Disease Control Over 36 Months
Description: Proportion of disease-free days in Step 2 or less (per Patient) using total number of days in study as the denominator- double-blind phase. Intent to Treat Population: defined as all randomized patients who were dispensed study medication and had at least one post baseline efficacy measurement.
Time Frame: 36 months
Population: Intent to Treat Population: all randomized patients who were dispensed study medication and had at least one post baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Proportion of disease free days
Arm/Group | Pimecrolimus (Elidel) Treatment Group | Control Treatment Group
Number analyzed (Participants) | 530 | 523
Proportion of disease free days | 0.4404 (0.29876) | 0.4346 (0.29317)
Statistical Analysis 1: Comparison: Pimecrolimus (Elidel) Treatment Group vs Control Treatment Group; A disease-free day in Step 2 or less was defined as a diary day with variable "No or almost no eczema?"=yes and "medication used variable"=no except emollients, yellow label medication 2X day, or medication deviation of yellow label medication 1x day; Test type: Superiority or Other; p = 0.7901, ANCOVA; Treatment, Center, gender, baseline age (months), baseline EASI score, and baseline TBSA as explanatory variables; Mean Difference (Final Values) = 0.0046, 95% CI 2-sided [-0.0290 to 0.0381]

2. Primary Outcome: Effect of Early Use of Pimecrolimus Cream 1% in Reducing the Incidence of Asthma at 6 Years of Age
Description: Note: The results for this efficacy variable are not reported due to early termination of the study.
Time Frame: 6 years
Reporting Status: Not Posted

3. Secondary Outcome: Long Term Safety in Infants and Young Children
Description: Note: The results of this secondary outcome is not reported due to early termination of the study.
Time Frame: 6 years
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Allergic Rhinitis, Allergic Conjunctivitis and Food Allergies
Description: Percentage of Patients who had allergic rhinitis, allergic conjunctivitis and food allergies at the end of the 36 month double blind study.
  Note: The results at six years are not reported due to early termination of the study.
Time Frame: 6 years (36 month Double-Blind Phase)
Population: Intent to Treat Population defined as all randomized patients who were dispensed study medication and had at least one post-baseline efficacy measurement.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pimecrolimus (Elidel) Treatment Group | Control Treatment Group
Number analyzed (Participants) | 533 | 532
Percentage of Participants
  Diagnosis of Food Allergy | 16.1 | 13.2
  Diagnosis of Allergic rhinitis | 18.6 | 16.4
  Diagnosis of Allergic conjunctivitis | 12.4 | 10.5

5. Secondary Outcome: Corticosteroid and Pimecrolimus Drug Use
Description: Corticosteroid and pimecrolimus study medication days of exposure during the 36 month double-blind phase.
  Note: Although the double-blind phase was designed to be 36 months (3 years) in length, the last double-blind visit for some patients occurred after 36 months.
Time Frame: 48 months
Population: Safety population: all randomized patients who were dispensed study medication.
Measure: Mean (Standard Deviation); unit: Days of Exposure
Arm/Group | Pimecrolimus (Elidel) Treatment Group | Control Treatment Group
Number analyzed (Participants) | 530 | 523
Days of Exposure
  Double -blind phase | 264.8 (259.49) | 249.6 (251.71)
  0-12 months (Year 1) | 146.6 (105.75) | 147.6 (112.69)
  13-24 months (Year 2) | 75.0 (105.08) | 65.0 (97.42)
  25-36 months (Year 3) | 42.2 (83.65) | 36.6 (76.31)
  37-48 months (Year 4) | 1.1 (5.74) | 1.0 (5.34)

6. Secondary Outcome: Atopic Dermatitis (AD) Remission Time
Description: Longest duration of atopic dermatitis (AD) remission during the 36 month double-blind treatment phase. A remission day was defined as a diary day with a positive response ("yes") to the question "No or almost no eczema?" and a response of no treatment except emollients to the question "Medication used".
Time Frame: 36 month Double-Blind Phase
Population: Intent-to-Treat population: all randomized patients who were dispensed study medication and had at least one post baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Pimecrolimus (Elidel) Treatment Group | Control Treatment Group
Number analyzed (Participants) | 530 | 523
Days | 105.9547 (137.61350) | 117.1071 (150.33993)

7. Secondary Outcome: Patient/Caregiver Quality of Life
Description: Change from Baseline in the total Parents' Index of Quality of Life-Atopic Dermatitis (PIQoL-AD) score in the double-blind phase. PIQoL-AD Score = (sum of valid items/number of valid items) * 28. Scores range from a minimum value of 0 to a maximum value of 28 with a high total overall score indicating poor quality of life.
Time Frame: From Baseline to Visit 5 , 6, 8, 10, 12, and 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on PIQoL-AD Scale
Arm/Group | Pimecrolimus (Elidel) Treatment Group | Control Treatment Group
Number analyzed (Participants) | 533 | 523
Scores on PIQoL-AD Scale
  Change in Baseline to Visit 5 (Week 14) | -2.6 (3.67) | -2.3 (3.37)
  Change in Baseline to Visit 6 (Week 27) | -2.7 (3.84) | -2.7 (3.83)
  Change in Baseline to Visit 8 (Week 53) | -2.9 (3.97) | -3.1 (4.23)
  Change in Baseline to Visit 10 (Week 88) | -3.1 (4.13) | -3.5 (4.23)
  Change in Baseline to Visit 12 (Week 122) | -3.3 (4.15) | -3.6 (4.39)
  Change in Baseline to Visit 14 (Week 158) | -3.5 (4.28) | -3.8 (4.35)

ADVERSE EVENTS:
Arm/Group | Pimecrolimus (Elidel) Treatment Group | Control Treatment Group
Serious Adverse Events (participants affected / at risk) | 42/543 | 37/544
Other Adverse Events (participants affected / at risk) | 482/543 | 467/544
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimecrolimus (Elidel) Treatment Group (N=543) | Control Treatment Group (N=544)
Pneumonia (Infections and infestations) | 6 | 6
Gastroenteritis rotavirus (Infections and infestations) | 3 | 4
Bronchiolitis (Infections and infestations) | 2 | 3
Gastroenteritis (Infections and infestations) | 2 | 2
Respiratory syncytial virus infection (Infections and infestations) | 2 | 2
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 2
Adenovirus infection (Infections and infestations) | 1 | 0
Croup, infectious (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Lymph node abscess (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Tonsillitis, streptococcal (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Beta hemolytic streptococcal infection (Infections and infestations) | 0 | 1
Eczema, infected (Infections and infestations) | 0 | 1
Laryngotracheo bronchitis (Infections and infestations) | 0 | 1
Pneumonia, bacterial (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Bronchial hyper-reactivity (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epiglottic edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 5
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 2
Food Allergy (Immune system disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 1 | 0
Milk allergy (Immune system disorders) | 0 | 1
Febrile convulsions (Nervous system disorders) | 2 | 2
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hepatic trauma (Injury, poisoning and procedural complications) | 0 | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Von Willebrand's disease (Congenital, familial and genetic disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nephroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Prepuce redundant (Reproductive system and breast disorders) | 1 | 0
Retinal hemorrhage (Eye disorders) | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pimecrolimus (Elidel) Treatment Group (N=543) | Control Treatment Group (N=544)
Upper Respiratory Tract Infection (Infections and infestations) | 288 | 265
Otitis Media (Infections and infestations) | 264 | 260
Nasopharyngitis (Infections and infestations) | 186 | 175
Gastroenteritis (Infections and infestations) | 76 | 69
Sinusitis (Infections and infestations) | 75 | 61
Gastroenteritis (Infections and infestations) | 55 | 50
Rhinitis (Infections and infestations) | 52 | 49
Croup infectious (Infections and infestations) | 46 | 51
Pharyngitis streptococcal (Infections and infestations) | 35 | 55
Pneumonia (Infections and infestations) | 45 | 44
Conjunctivitis, bacterial (Infections and infestations) | 39 | 45
Viral upper respiratory tract infection (Infections and infestations) | 37 | 38
Bronchitis (Infections and infestations) | 41 | 30
Bronchiolitis (Infections and infestations) | 28 | 33
Impetigo (Infections and infestations) | 22 | 37
Viral rash (Infections and infestations) | 29 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 187 | 174
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 122 | 107
Wheezing (Respiratory, thoracic and mediastinal disorders) | 102 | 89
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 68 | 63
Asthma (Respiratory, thoracic and mediastinal disorders) | 64 | 53
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 52 | 43
Diarrhea (Gastrointestinal disorders) | 55 | 46
Teething (Gastrointestinal disorders) | 134 | 135
Vomiting (Gastrointestinal disorders) | 34 | 29
Food Allergy (Immune system disorders) | 140 | 118
Milk allergy (Immune system disorders) | 50 | 35
Pyrexia (General disorders) | 123 | 123
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 44 | 46
Urticaria (Skin and subcutaneous tissue disorders) | 41 | 31
Conjunctivitis, allergic (Eye disorders) | 76 | 63
Conjunctivitis (Eye disorders) | 50 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.